CLINICAL TRIAL: NCT02831881
Title: PROTECTED PCI STUDY: A Prospective Clinical Trial For Patients Undergoing Protected Percutaneous Coronary Intervention With IMPELLA® 2.5 System
Brief Title: Protected PCI Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abiomed Inc. (Industry)
Collaborators: Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Other Study IDs: PROTECT III
Record Dates: First submitted 2016-07-01; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A Prospective, multi-center, single-arm post-approval study of the IMPELLA® 2.5 System in Non Emergent High Risk PCI patients.

DETAILED DESCRIPTION:
The objective of the study is to assess the safety and efficacy of the IMPELLA® 2.5 System in subjects undergoing non-emergent high-risk percutaneous coronary intervention (PCI) post market approval. The primary endpoint will be a composite clinical endpoint of major adverse events through 90 days following the PCI procedure. The outcome will be compared to the pre specified performance goal of 53%.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Subject is indicated for a NON emergent percutaneous treatment of at least one de novo or restenotic lesion in a native coronary vessel or bypass graft per the judgement of a heart team including a surgeon
3. Age eligible (18 ≤ Age ≤ 90)
4. Subject presents with:

   1. Ejection Fraction≤ 35% AND at least one of the following criteria:

      Intervention on the last patent coronary conduit, or Intervention on an unprotected left main coronary artery Or
   2. Ejection Fraction ≤ 30% and intervention in patient presenting with triple vessel disease. *three-vessel or triple vessel disease is defined as at least one significant stenosis* in all three major epicardial territories: Left Anterior Descending (LAD) Artery and/or side branch, left circumflex (LCX) artery and/or side branch, Right Coronary Artery (RCA) and or side branch. *Significant stenosis is defined as at least 50% diameter stenosis by visual estimate or any total occlusion. In the case of left coronary artery dominance, a lesion in the LAD and the proximal LCX qualifies as three-vessel disease.

Exclusion Criteria:

* 1. ST Myocardial Infarction within 24 hours or CK-MB that have not normalized

  2. Pre-procedure cardiac arrest within 24 hours of enrolment requiring CPR

  3. Subject is inotrope dependent or in cardiogenic shock defined as: Hypotension (systolic BP < 90 mmHg for > 30 minutes or the need for supportive measures to maintain a systolic BP of greater than or equal to 90 mmHg) AND end organ hypoperfusion (cool extremities OR a urine output of < 30 ml/hour)

  4. Mural thrombus in the left ventricle

  5. Patient scheduled for revascularization of a total chronic occlusion (CTO) or transcatheter aortic valve replacement within 1 year of index procedure.

  6. The presence of a mechanical aortic valve or heart constrictive device

  7. Documented presence of aortic stenosis (aortic stenosis graded as ≥ +2 equivalent to an orifice area of 1.5cm2 or less.

  8. Documented presence of moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as ≥ +2)

  9. Severe peripheral arterial obstructive disease that would preclude the IMPELLA System device placement

  10. Abnormalities of the aorta that would preclude surgery, including aneurysms and extreme tortuosity or calcifications

  11. Subject with renal failure (creatinine ≥ 4mg/dL or on dialysis)

  12. Subject has history of debilitating liver dysfunction with elevation of liver enzymes and bilirubin levels to ≥ 3x ULN or INR (Internationalized Normalized Ratio) ≥ 2

  13. Subject has uncorrectable abnormal coagulation parameters (defined as platelet count ≤75,000/mm3 or INR ≥2.0.)

  14. History of recent (within 1 month) stroke or TIA

  15. Allergy or intolerance to heparin, aspirin, ADP receptor inhibitors(clopidogrel and ticlid) or contrast media

  16. Subject with documented heparin induced thrombocytopenia

  17. Participation in the active follow-up phase of another clinical study of an investigational drug or device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of high risk subjects indicated for nonemergent percutaneous treatment after heart team evaluation including a cardiac surgeon of at least one de novo or restenotic lesion in a native coronary vessel or bypass graft.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
A composite rate of the following intra-procedural and post-procedural major adverse events (MAE) at 90 days post index procedure. | 90 days post index procedure
  The primary endpoint is defined as a composite rate of the major adverse events at 90 days post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided